CLINICAL TRIAL: NCT00048360
Title: An 8-week, Multicenter, Randomized, Double-Blind, Placebo-Controlled, Flexible-Dose Comparison of Extended-Release Bupropion Hydrochloride 300-450 mg/Day to Assess the Efficacy, Safety, and Effects on Health Outcomes in the Treatment of Adults With Attention-Deficit/Hyperactivity Disorder
Brief Title: Attention-Deficit Hyperactivity Disorder (ADHD) Study With Adults
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AK130934
Record Dates: First submitted 2002-10-30; First posted 2002-10-31 (Estimated); Last update posted 2013-02-12 (Estimated); Status verified 2013-02

CONDITIONS: Attention Deficit Disorder
Keywords: ADD; ADHD; attention deficit; hyperactivity
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Spasm

INTERVENTIONS:
Drug: Extended-release bupropion hydrochloride

SUMMARY:
This is a placebo controlled study evaluating the efficacy and safety of medication in adults with Attention-Deficit Hyperactivity Disorder (ADHD).

ELIGIBILITY:
Inclusion criteria:

* Patient must be diagnosed with ADHD.

Exclusion Criteria:

* Patient has a current or past history of seizure disorder, brain injury, anorexia nervosa or bulimia.
* Patient has a current diagnosis of Major Depressive Disorder (MDD).
* Patient has a current primary diagnosis of, or received treatment for, Panic Disorder, Obsessive Compulsive Disorder (OCD), Posttraumatic Stress Disorder (PTSD) or Acute Stress Disorder within the previous 12 months.
* Patient has a lifetime diagnosis of bipolar disorder, schizophrenia or other psychotic disorders.
* Patient has a positive urine test at screening for presence of illicit drugs or alcohol abuse during the past 12 months.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 162
Dates: Start 2002-10; Primary Completion 2003-06 (Actual); Study Completion 2003-06 (Actual)

PRIMARY OUTCOMES:
ADHD Rating Scale

SECONDARY OUTCOMES:
Clinical Global Impressions -Severity and Improvement.
Quality of Life Enjoyment and Satisfaction Questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trial, MD, Study Chair — GlaxoSmithKline
Locations (21):
- United States (21):
  - GSK Clinical Trials Call Center, Phoenix, Arizona
  - GSK Clinical Trials Call Center, Chula Vista, California
  - GSK Clinical Trials Call Center, Lafayette, California
  - GSK Clinical Trials Call Center, Northridge, California
  - GSK Clinical Trials Call Center, Spring Valley, California
  - GSK Clinical Trials Call Center, West Palm Beach, Florida
  - GSK Clinical Trials Call Center, Paducah, Kentucky
  - GSK Clinical Trials Call Center, Rockville, Maryland
  - GSK Clinical Trials Call Center, Cambridge, Massachusetts
  - GSK Clinical Trials Call Center, Worcester, Massachusetts
  - GSK Clinical Trials Call Center, Omaha, Nebraska
  - GSK Clinical Trials Call Center, Chapel Hill, North Carolina
  - GSK Clinical Trials Call Center, Beachwood, Ohio
  - GSK Clinical Trials Call Center, Cincinnati, Ohio
  - GSK Clinical Trials Call Center, Portland, Oregon
  - GSK Clinical Trials Call Center, Bellaire, Texas
  - GSK Clinical Trials Call Center, Houston, Texas
  - GSK Clinical Trials Call Center, Salt Lake City, Utah
  - GSK Clinical Trials Call Center, Burlington, Vermont
  - GSK Clinical Trials Call Center, Woodstock, Vermont
  - GSK Clinical Trials Call Center, Seattle, Washington